CLINICAL TRIAL: NCT06705842
Title: The APPI-Cost Trial: Cost Assessment of Povidone-Iodine Irrigation for Prevention of Intra-abdominal Abscess in Perforated Appendicitis
Brief Title: APPI-Cost Trial for Perforated Appendicitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Dalya M Ferguson, MD, MS, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-24-0772; 1K12TR004908-01 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Perforated Appendicitis
Keywords: Perforated Appendicitis; Povidone Iodine; Cost effectiveness; Intra-abdominal abscess; Appendectomy; Implementation science
MeSH Terms: conditions — Appendicitis; Abdominal Abscess

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PVI (Active Comparator)
  Interventions: Drug: PVI
- Usual Care (Active Comparator)
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: PVI — After removal of the appendix from the patient's abdomen and attainment of hemostasis, 10 mL/kg of 1% PVI (up to a maximum of 1,000 mL) will be used to irrigate the pelvis and right upper and lower quadrants. The solution will be left to dwell for 1 minute and then suctioned out
  Arms: PVI
Drug: Usual Care — Surgeons may utilize local irrigation with saline if deemed necessary, defined as instillation of a small volume (<100 mL) of liquid followed by aspiration, for the purpose of confirming hemostasis or suctioning thick fluid. Some surgeons may utilize large volume irrigation with saline solution, if that is consistent with their usual practice. Patients in the usual care arm will not receive PVI irrigation.
  Arms: Usual Care

SUMMARY:
The purpose of this study to assess the clinical effectiveness and cost-effectiveness of povidone-iodine (PVI) irrigation in perforated appendicitis, to investigate barriers and facilitators to future implementation of PVI irrigation, and to collect costs and clinical and patient-reported outcomes among patients with non-perforated appendicitis.

ELIGIBILITY:
Eligibility for Enrollment

Inclusion Criteria:

* Plan to undergo appendectomy for acute appendicitis

Exclusion Criteria:

* Preoperative hemodynamic instability requiring ongoing infusion of vasopressors
* Allergy to iodine
* Uncontrolled hyper- or hypothyroidism
* Renal dysfunction
* Pregnant or breastfeeding
* Primary language neither English nor Spanish
* Lack of functioning telephone or email account
* Incarcerated or in police custody

Eligibility for Randomization

Inclusion Criteria:

* Enrolled in study preoperatively
* Intraoperative diagnosis of perforated appendicitis

Exclusion Criteria:

* Non-perforated appendicitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness of PVI relative to usual care | 30 day follow up
  Cost-effectiveness of PVI irrigation relative to usual care will be assessed as the incremental 30-day total societal costs per percent reduction in IAA rate. The Incremental Cost Effectiveness Ratio (ICER) will be calculated as: (societal costs with PVI irrigation minus societal costs with usual care) divided by (IAA rate with PVI minus IAA rate with usual care). IAA will be defined as an image-confirmed fluid collection deemed to be an IAA by an attending surgeon or radiologist, or an abscess confirmed during percutaneous intervention or reoperation. Societal costs will be defined as patient-reported costs plus medical costs for inpatient and outpatient care within 30 days from randomization. PVI will be deemed cost-effective by either 1) reducing 30-day IAA rate without increasing 30-day total societal costs, 2) reducing 30-day total societal costs without increasing 30-day IAA rate, or 3) reducing both 30-day societal costs and IAA rate.

SECONDARY OUTCOMES:
Total patient-reported costs | 30 days, 90 days, 6 months, and 12 months
  Patient-reported costs will be assessed using a patient survey, which will be verbally administered by research personnel at each time point specified.
Health-related quality of life as assessed by the EQ-5D-5L questionnaire | 30 days, 90 days, 6 months, and 12 months
  This is a 6 item questionnaire and the first 5 questions are each scored from 1 (no problem) - 5 (unable to), for a maximum score of 25, with a higher number indicating a worse outcome. The 6th question is scored on a Likert scale from 0 (worst health you can imagine) - 100 (best health you can imagine), with a higher score indicating a worse outcome.
Index admission total hospital costs | Index admission (variable duration)
90-day total hospital costs | 90 day follow up
Index admission total length of hospital stay | Index admission (variable duration)
90-day total length of hospital stay | 90 day follow up
Number of days of work missed by participant | 12 months
Postoperative complications | 90 days follow up
  Complications include IAA, clinically relevant IAA, superficial/deep surgical site infection, ED visit, readmission, reoperation, subsequent procedure, or mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dalya Ferguson, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Starting 6 months after study publication, de-identified data and study materials may be made available to researchers on a case-by-case basis.